CLINICAL TRIAL: NCT04249310
Title: Early Intervention Effectiveness of Tiotropium / Olodaterol Compared to Tiotropium in COPD
Brief Title: Early Intervention Efficacy in COPD
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0100
Record Dates: First submitted 2020-01-29; First posted 2020-01-30 (Actual); Results first posted 2021-08-30 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol; Tiotropium Bromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes

GROUPS / COHORTS (2):
- Tiotropium/Olodaterol: Combination of Tiotropium and Olodaterol
  Interventions: Drug: Tiotropium/Olodaterol
- Tiotropium
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: Tiotropium/Olodaterol — Soft Mist Inhaler product
  Other Names: Spiolto®
  Groups: Tiotropium/Olodaterol
Drug: Tiotropium — Soft Mist Inhaler product
  Other Names: Spiriva®
  Groups: Tiotropium

SUMMARY:
This study aims to evaluate the time to escalation to triple therapy among the Japanese Chronic obstructive pulmonary disease (COPD) patients newly initiating therapy with a combination of Olodaterol and Tiotropium (herein referred to as Tio/Olo) using real world data.

ELIGIBILITY:
Inclusion Criteria:

The study cohort will include all patients who initiate Tiotropium/ Olodaterol (Tio/Olo) or Tiotropium (Tio) during the patient selection period.

Exclusion Criteria:

The following exclusion criteria will then be applied to generate the unmatched cohort:

* Aged <40 years on cohort entry.
* Any LAMA, LABA, or ICS maintenance therapy (alone or in combination) during the 180-day baseline period prior to cohort entry for maintenance treatment and duration >30 days, or any prescription within the 30 days prior to cohort entry.
* Patients without continuous enrolment (days since first inpatient/ outpatient encounter in the data) during the baseline period.
* No prior diagnosis of COPD [International Classification of Diseases (ICD)-10: J41*, J43*, J44* and doubt (UTAGAIFLG) = 0 (no)]
* Patients without a second prescription claim of their index medication within 60 days after the cohort entry date.
* Diagnosis of asthma [ICD-10: J45* and doubt (UTAGAIFLG) = 0 (no)] during the baseline period.
* Diagnosis of lung cancer [ICD-10: C34*, D02.2, Z80.1, Z85.1 and doubt (UTALAIFLG) = 0 (no)] or lung transplant (Health claim code: 150317670, 150322510, 150322610, 150336510, 150336610, 150336710, 150399270) prior to the cohort entry date using all available data.
* Patients who initiate both Tio/Olo and Tio simultaneously on the cohort entry date.
* Any use of triple therapy (LAMA + LABA + ICS) during the baseline period or between the cohort entry date and 1 day prior to the start of follow-up.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort will include all patients who initiate Tiotropium/Olodaterol (Tio/Olo) or Tiotropium (Tio) during the patient selection period. Initiation (new use) will be determined based on no prescription claims for Tio/Olo or Tio during the baseline period or during all available data prior to cohort entry date. All patients will additionally be required to have a second claim for the index medication within 60 days after cohort entry to ensure primary adherence of index therapy.
Sampling Method: Probability Sample
Enrollment: 6788 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nara Medical University, Nara, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A new-user, active comparator retrospective comparative cohort study using a Japanese electronic healthcare research database.The study aims to test early intervention effectiveness of tiotropium/olodaterol compared to tiotropium in patients with chronic obstructive pulmonary disease (COPD).
Pre-assignment Details: Only subjects that met all inclusion and none of the exclusion criteria were included in the study. The enrolled patients were matched into 2 (not mutually exclusive) cohorts: 1) basic propensity score (PS) cohort, 2) high dimensional propensity score (hdPS) cohort.
Groups:
- Tiotropium/Olodaterol (Spiolto®): All patients with chronic obstructive pulmonary disease (COPD), included in the Japanese electronic healthcare research database (MDV Japan), who initiated Tiotropium/Olodaterol (Tio/Olo) during the patient selection period (September 2015 to December 2018). Patients were followed up a maximum of 360 days or until end of study period (March 2019, end of available data).
- Tiotropium (Spiriva®): All patients with chronic obstructive pulmonary disease (COPD), included in the Japanese electronic healthcare research database (MDV Japan), who initiated Tiotropium during the patient selection period (September 2015 to December 2018). Patients were followed up a maximum of 360 days or until end of study period (March 2019, end of available data).
Period: Overall Study
Arm/Group | Tiotropium/Olodaterol (Spiolto®) | Tiotropium (Spiriva®)
Started (Unmatched cohort) | 1436 | 5352
PS-matched Cohort | 1412 | 1412
hdPS-matched Cohort | 1302 | 1302
Completed | 1436 | 5352
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients included on the Japanese electronic, record based health care database (MDV) between September 2015 and December 2019 using either a combination of tiotropium/olodaterol or tiotropium alone - unmatched cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium/Olodaterol (Spiolto®) | Tiotropium (Spiriva®) | Total
Number analyzed (Participants) | 1436 | 5352 | 6788
Age, Continuous [Mean (Standard Deviation); unit: Years] — All patients included on the Japanese electronic, record based health care database (MDV) between September 2015 and December 2019 using either a combination of tiotropium/olodaterol or tiotropium alone - unmatched cohort.
  Years | 75.16 (8.41) | 75.56 (8.90) | 75.48 (8.80)
Sex: Female, Male [Count of Participants; unit: Participants] — All patients included on the Japanese electronic, record based health care database (MDV) between September 2015 and December 2019 using either a combination of tiotropium/olodaterol or tiotropium alone - unmatched cohort.
  Participants
    Female | 163 | 779 | 942
    Male | 1273 | 4573 | 5846
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time to Triple Therapy Initiation
Description: Time to triple therapy initiation (first event per patient) defined as any fixed dose combination of Long-acting muscarinic antagonists (LAMA) / Long-acting beta agonist (LABA) / Inhaled Corticosteroid (ICS) or any concurrent use for 30 consecutive days of the following:
  * any LAMA/LABA fixed dose combination + any ICS single formulation
  * any LAMA single formulation + any LABA/ICS fixed dose combination
  * any LAMA single formulation + any LABA single formulation + any ICS single formulation.
  Patients will be censored if they had an occurrence of any of the following: outcome (initiation of triple therapy), death, or end of data. The analysis will use an intention-to-treat censoring approach, which does not account for treatment change.
Time Frame: From index date (cohort entry date) until first occurence of event, up to 42 months.
Population: All patients included on the Japanese electronic, record based health care database (MDV) between September 2015 and December 2019 using either a combination of tiotropium/olodaterol or tiotropium alone - High dimensional propensity score (hdPS) matched cohort.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Tiotropium/Olodaterol (Spiolto®) | Tiotropium (Spiriva®)
Number analyzed (Participants) | 1302 | 1302
Days | 195.0 (123.2) | 89.5 (112.3)
Statistical Analysis 1: Comparison: Tiotropium/Olodaterol (Spiolto®) vs Tiotropium (Spiriva®); Test type: Other; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.32 to 2.46] — [(Tiotropium/Olodaterol) / Tiotropium] Cox-regression was used to estimate the hazard ratios and 95% confidence intervals

2. Secondary Outcome: Time to First Moderate or Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Description: Time to First Moderate or Severe COPD Exacerbation. Moderate exacerbation is defined as an outpatient visit with a diagnosed code for COPD in any field + a prescription for an oral corticosteroid or an antibiotic for respiratory infections. Severe exacerbations will be defined as a hospitalization with a primary diagnosis for COPD.
  Patients will be censored if they had an occurrence of any of the following: outcome (initiation of triple therapy), death, or end of data. The analysis will use an intention-to-treat censoring approach, which does not account for treatment change.
Time Frame: From index date until first occurence of event, up to 42 months.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Tiotropium/Olodaterol (Spiolto®) | Tiotropium (Spiriva®)
Number analyzed (Participants) | 1302 | 1302
Days
  Moderate or Severe | 116.3 (108.7) | 118.8 (105.9)
  Moderate Exacerbation | 125.6 (107.4) | 139.0 (121.3)
  Severe Exacerbation | 134.0 (112.5) | 134.5 (107.1)
Statistical Analysis 1: Comparison: Tiotropium/Olodaterol (Spiolto®) vs Tiotropium (Spiriva®); Moderate or Severe COPD Exacerbation; Test type: Other; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.63 to 1.15] — [(Tiotropium/Olodaterol) / Tiotropium] Cox regression was used to estimate the hazard ratios and 95% confidence intervals
Statistical Analysis 2: Comparison: Tiotropium/Olodaterol (Spiolto®) vs Tiotropium (Spiriva®); Moderate COPD Exacerbation; Test type: Other; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.43 to 1.01] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Tiotropium/Olodaterol (Spiolto®) vs Tiotropium (Spiriva®); Severe COPD Exacerbation; Test type: Other; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.62 to 1.31] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Number of Moderate or Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbations
Description: Number of Moderate or Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbations.
  Moderate exacerbation is defined as an outpatient visit with a diagnosed code for COPD in any field + a prescription for an oral corticosteroid or an antibiotic for respiratory infections. Severe exacerbations will be defined as a hospitalization with a primary diagnosis for COPD.
  Patients will be censored if they had an occurrence of any of the following: outcome (initiation of triple therapy), death, or end of data. The analysis will use an intention-to-treat censoring approach, which does not account for treatment change.
Time Frame: From index date until first occurence of event, up to 42 months.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Number of Exacerbations
Arm/Group | Tiotropium/Olodaterol (Spiolto®) | Tiotropium (Spiriva®)
Number analyzed (Participants) | 1436 | 5352
Number of Exacerbations
  Moderate or Severe Exacerbations | 0.08 (0.33) | 0.08 (0.34)
  Moderate Exacerbations | 0.04 (0.22) | 0.04 (0.22)
  Severe Exacerbations | 0.05 (0.24) | 0.05 (0.27)

ADVERSE EVENTS:
Description: As this is a non-interventional study with secondary use of data retrieved from a Japanese database, safety monitoring and safety reporting on an individual case level is not applicable. All-Cause Mortality, Serious Adverse Events and Other Adverse Events are not collected in the database. "0" total Number of Participants at Risk means "All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed".
Arm/Group | Tiotropium/Olodaterol (Spiolto®) | Tiotropium (Spiriva®)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT04249310/Prot_SAP_000.pdf